CLINICAL TRIAL: NCT00999882
Title: A Phase I/II, Open-label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Tor Kinase Inhibitor (AZD8055) in Asian Patients With Advanced Stage Hepatocellular Carcinoma (HCC) and With Mild or Moderate Hepatic Impairment
Brief Title: Safety, Tolerability, Pharmacokinetics (PK) and Preliminary Efficacy of Tor Kinase Inhibitor in Liver Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1600C00014
Record Dates: First submitted 2009-10-13; First posted 2009-10-22 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Cancer; Advanced Hepatocellular Carcinoma
Keywords: mTor Kinase Inhibitor; Phase I/II; Dose escalation; Hepatocellular carcinoma (HCC); Asia; HCC; Safety and pharmacokinetics
MeSH Terms: conditions — Neoplasms; Carcinoma, Hepatocellular | interventions — (5-(2,4-bis((3S)-3-methylmorpholin-4-yl)pyrido(2,3-d)pyrimidin-7-yl)-2-methoxyphenyl)methanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZD8055 (Experimental): Dose escalation
  Interventions: Drug: AZD8055

INTERVENTIONS:
Drug: AZD8055 — Dose escalation phase: Tablet taken orally, a single dose of AZD8055 on Day 1, followed by twice daily continuous dosing from Day 3 onwards, till discontinuation or withdrawal.Expansion phase: twice daily continuous dosing from Day 1 onwards till discontinuation or withdrawal.

SUMMARY:
The main purpose of the study is to establish a safe dose of AZD8055 in patients with mild or moderate liver disease by providing information on any potential side effects this drug may cause and collecting data about how hepatocellular carcinoma responds to the drug.

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage Hepatocellular Carcinoma (HCC) confirmed by cytology or histology
* Advanced stage Hepatocellular Carcinoma (HCC) or metastatic Hepatocellular Carcinoma (HCC) which is inoperable and incurable with standard available treatments
* Relatively good overall health other than cancer (WHO performance status (0-2)

Exclusion Criteria:

* Patients with severe heart conditions, or those who have had heart surgery such as coronary artery bypass graft within the last 6 months, or patients with uncontrolled high blood pressure despite medical management.
* Patients must not have received any other anti cancer therapy including TACE within 21 days of entering the trial
* Patients must not have received a liver transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability (Adverse events, vital signs, ECG, chemistry, haematology, urinalysis, physical examination) | Every week for Cycle 1 and 2, every 2 weeks from cycle 3 onwards, every 4 weeks from cycle 7 onwards
Evaluate the pharmacokinetics of AZD8055 following both single and multiple dosing | Blood samples on 6 occasions during the first Cycle of the study (28 days)

SECONDARY OUTCOMES:
To make a preliminary assessment of efficacy | Every 4 weeks
To investigate the possible relationship between plasma concentration of AZD8055 concentrations and the extent of liver impairment. | During Cycle 1 of the study - blood samples before study treatment and then on Day 1, 3, 10, 17, 24, 30 and then on day 1 of every cycle
Evaluate the change in Phosphorylation levels of certain biomarkers before and after treatment with AZD8055 | Blood samples x 3 times on Day 1 of the first cycle
To collect and store DNA for future exploratory research that may influence response to AZD8055 | Blood sample on Day 1 or at any other visit during study
  May not be reported in the CSR

CONTACTS AND LOCATIONS:
Overall Officials: Brigette Ma, Principal Investigator — Prince of Wales Hospital, HongKong; Ian Smith, Study Director — AstraZeneca
Locations (3):
- Research Site, Hong Kong, Hong Kong
- South Korea (2):
  - Research Site, Seongnam-si, Gyeonggi-do
  - Research Site, Seoul